CLINICAL TRIAL: NCT01496781
Title: EndoClotTM Absorbable Polysaccharide Hemostat in Comparison With Metallic Hemoclip for Hemostasis and Preventing Post-procedure Bleeding After Endoscopic Mucosal Resection: a Prospective, Randomized Trial
Brief Title: EndoClot for Hemostasis and Preventing Post-procedure Bleeding After Endoscopic Mucosal Resection
Acronym: EMR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Zhiguo Liu, Associated Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20111219
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Endoscopic Hemostasis; Colonic Polyps
Keywords: Endoscopic Hemostasis; metallic hemoclip; EndoClot Absorbable Polysaccharide Hemostat; Colonic Polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EndoClot (Experimental): This arm is designed to observe if the Endoclot treatment can achieve comparable hemostasis efficacy compared with hemoclip.
  Interventions: Procedure: EndoClot
- Hemoclip (Active Comparator): This arm is used as a control treatment group to compare with Endoclot treatment.
  Interventions: Procedure: Hemoclip

INTERVENTIONS:
Procedure: Hemoclip — Hemoclip application is a standard treatment option after endoscopic mucosal resection of colonic lesion to stop and prevent post-procedure bleeding.
  Other Names: metallic hemoclip (Cat# HX-610-090L, Olympus)
  Arms: Hemoclip
Procedure: EndoClot — EndoClot hemostat is applied immediately after EMR to achieve hemostasis.
  Other Names: EndoClot® Absorbable Polysaccharide Hemostat (Cat# Y2007090722, Starch Medical Inc)
  Arms: EndoClot

SUMMARY:
Endoscopic mucosal resection (EMR) has been widely used as a diagnostic and treatment techniques of gastrointestinal small lesions. Para-procedure bleeding is one of the common complication following EMR. Several endoscopic hemostasis methods are currently in use including metallic hemoclip. EndoClot® absorbable polysaccharide hemostat (PAPH) as a new hemostasis material was previously used for surgical hemostasis, but the therapeutic effect and safety in endoscopic application remains unknown. This randomized controlled study has been designed to compare PAPH with metallic hemoclip in their hemostatic effect of intra-procedure bleeding control and rebleeding prevention during and after EMR.

ELIGIBILITY:
Inclusion Criteria:

* consecutive cases of colorectal polyps and submucosal tumors with anticipated complete removal endoscopically by EMR.

Exclusion Criteria:

* severe cardiovascular diseases, liver and kidney dysfunction;
* platelet and coagulation dysfunction (PLT < 50*109/L, INR > 2);
* cases that have taken anticoagulant drugs or non-steroidal anti-inflammatory drugs within 1 month before the procedure;
* cases unavailable for follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2010-04; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Hemostasis rate after EMR | Up to half an hour immediately after EMR procedure to ensure successful management is achieved.
  Initial hemostatsis was observed endoscopically immediately after application of hemoclip or Endoclot. Complete hemostatsis is ensured. Endoscopic combined hemostasis or emergency surgery would be applied if severe bleeding occurred and endoscopic management fails

SECONDARY OUTCOMES:
Mucosal healing after EMR | up to 1 month
  Colonoscopy will be repeated 1 month after EMR procedure to observe if application of Endoclot will delay the musosal healing.
Time taken to achieve hemostasis | Up to half an hour immediately after EMR procedure to ensure successful management is achieved.
  The time taken to achieve hemostasis is recorded immediately after EMR procedure to reflect the technical difficulty of hemostasis measure.
Rebleeding rate after EMR procedure | up to 1 week
  Rebleeding rate up to 1 week was obtained by clinical manifestations such as melana; decreased hemoglobin > 20g/L; hemodynamic instability or active bleeding from mucosal defect under endoscope.
gastrointestinal tract obstruction | up to 1 month
  Gastrointestinal tract obstruction has been previously reported as a possible adverse effect of hemostats, therefore it was observed in the current study.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Parra-Blanco A, Kaminaga N, Kojima T, Endo Y, Uragami N, Okawa N, Hattori T, Takahashi H, Fujita R. Hemoclipping for postpolypectomy and postbiopsy colonic bleeding. Gastrointest Endosc. 2000 Jan;51(1):37-41. doi: 10.1016/s0016-5107(00)70384-1. PMID 10625793
- [Background] Lin LF, Siauw CP, Ho KS, Tung JC. Endoscopic hemoclip treatment of gastrointestinal bleeding. Chang Gung Med J. 2001 May;24(5):307-12. PMID 11480327
- [Background] Binmoeller KF, Thonke F, Soehendra N. Endoscopic hemoclip treatment for gastrointestinal bleeding. Endoscopy. 1993 Feb;25(2):167-70. doi: 10.1055/s-2007-1010277. PMID 8491134
- [Background] Katsinelos P, Paroutoglou G, Beltsis A, Papaziogas B, Gouvalas A, Chatzimavroudis G, Vlachakis I, Mimidis K, Vradelis S, Pilpilidis I. Endoscopic hemoclip application in the treatment of nonvariceal gastrointestinal bleeding: short-term and long-term benefits. Surg Laparosc Endosc Percutan Tech. 2005 Aug;15(4):187-90. doi: 10.1097/01.sle.0000174575.52840.23. PMID 16082303
- [Background] Kouklakis G, Mpoumponaris A, Gatopoulou A, Efraimidou E, Manolas K, Lirantzopoulos N. Endoscopic resection of large pedunculated colonic polyps and risk of postpolypectomy bleeding with adrenaline injection versus endoloop and hemoclip: a prospective, randomized study. Surg Endosc. 2009 Dec;23(12):2732-7. doi: 10.1007/s00464-009-0478-3. Epub 2009 May 9. PMID 19430833
- [Background] Wang Y, Xu M, Dong H, Liu Y, Zhao P, Niu W, Xu D, Ji X, Xing C, Lu D, Li Z. Effects of PerClot(R) on the healing of full-thickness skin wounds in rats. Acta Histochem. 2012 Jul;114(4):311-7. doi: 10.1016/j.acthis.2011.06.012. Epub 2011 Jul 22. PMID 21782216